CLINICAL TRIAL: NCT06580431
Title: Trimethylamine N-oxide (TMAO) Levels in Periodontal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Nur Balci, DDs, PhD, DDs, PhD, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1061
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Periodontitis; Smoking; Inflammatory Response
Keywords: periodontal disease; smoking; TMAO
MeSH Terms: conditions — Periodontitis; Smoking; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Saliva and serum of periodontitis and smoking patients collected for analyzing TMAO levels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): Saliva and serum collection of patients and samples molecules analysis Saliva and serum sampling Saliva were collected to analyze the selected markers as unstimulated samples during the early hours of the day. The saliva was centrifuged and then transferred into Eppendorf tubes. Venous puncture was performed after saliva collection and 10 mL of blood samples were collected by qualified staff from each participant. Saliva and serum were then stored at -80 °C until analysis.
  Interventions: Other: Saliva and serum sampling
- Salivary and serum TMAO observation (Experimental): TNF-α levels in collected saliva and serum samples were measured by commercial ELISA kits (ELISA Cloud Immunoassay, Cloud Clone Corp; cat #SEA079Hu) and analyzed according to manufacturers' instructions. The standard curve of the assay was used to determine the analyte concentrations in each sample. All samples were analyzed in duplicate, and the mean values were used in subsequent calculations.
  TMAO levels in saliva and serum were determined by a liquid chromatography-mass spectrometry (LC MS/MS) method (LC-MS/MS, ESI Source, Thermo Scientific Accessmax), which was a modification of the method by Li et al and similar as our previous study.(Yufei Li, Kang, Lee, Chung, & Cho, 2021) To identify and quantify TMAO, samples were analyzed by an LC-MS/MS 1 system equipped with a Thermo Dionex Ultimate 3000 UHPLC system and an TSQ Quantum Access Max quadrupole mass spectrometer (USA).
  Interventions: Other: Saliva and serum sampling

INTERVENTIONS:
Other: Saliva and serum sampling — Saliva were collected to analyze the selected markers as unstimulated samples during the early hours of the day. The saliva was centrifuged and then transferred into Eppendorf tubes. Venous puncture was performed after saliva collection and 10 mL of blood samples were collected by qualified staff from each participant. Saliva and serum were then stored at -80 °C until analysis.

SUMMARY:
Salivary and serum levels of TMAO and TNF-A can distinguish between individuals with periodontitis and periodontally healthy persons, including smoking and nonsmoking patients.

DETAILED DESCRIPTION:
Tobacco use is a prevalent global habit with notable impacts on general health and periodontal disease. Trimethylamine N-oxide (TMAO) is a compound involved in the pathogenesis of various systemic inflammatory diseases, including cardiovascular conditions. The aim of this study was to determine differences in saliva and serum levels of TMAO between periodontitis and periodontally healthy patients according to smoking status.

The study includes four groups: systemically and periodontally healthy non-smokers (NS- Control; n = 25), systemically healthy non-smokers with Stage-III Grade-B periodontitis (NS- Periodontitis; n = 25), systemically and periodontally healthy smokers (S-Control; n = 25), and systemically healthy smokers with Stage-III Grade-C periodontitis (S-Periodontitis; n = 25). Periodontal parameters were recorded. TMAO levels were determined in saliva and serum samples using liquid chromatography-mass spectrometry (LC-MS/MS). TNF-α levels were measured by ELISA method.

ELIGIBILITY:
Inclusion Criteria:

* • systemically healthy

  * clinical diagnosis of periodontitis
  * clinical diagnosis of periodontal health
  * For smoking group : denied as smoking at least 10 cigarettes per day and the duration should more than 10 years.

Exclusion Criteria:

* decline to participate and being under 18 & over 65 years of age; (2) having any systemic inflammatory diseases such as diabetes, rheumatoid arthritis, or systemic conditions, including immunodeficiency syndrome, cardiovascular disorders, or hepatic disorders; (3) the use of antibiotics and/or anti-inflammatory nonsteroidal anti-inflammatory drugs within 3 months preceding the study; (4) having nonsurgical periodontal treatment (previous 6 months); (5)having surgical periodontal treatment (previous 12 months); (6)having <20 natural teeth excluding the third molars.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Pocket probing depth | 3 months
  Measurement of the depth of a sulcus or periodontal pocket determined by measuring distance from a gingival margin to the base of the sulcus or pocket with a calibrated periodontal probe
Clinical attachment level | 4 months
  Clinical attachment level (or loss, CAL) is a more accurate indicator of the periodontal support around a tooth than probing depth alone. CAL is measured from a fixed point on the tooth that does not change, the CEJ.
  To calculate CAL, two measurements are needed: distance from the gingival margin to the CEJ and probing depth.
  In recession: probing depth (+) gingival margin to the CEJ (add). In tissue overgrowth: probing depth (-) gingival margin to the CEJ (subtract)
Bleeding on probing | 4 months
  Bleeding on probing referring to bleeding that is induced by gentle manipulation of the tissue at the depth of the gingival sulcus, or interface between the gingiva and a tooth

SECONDARY OUTCOMES:
serum and saliva analyses for TMAO levels | 1 month
  TMAO levels were determined in saliva and serum samples using liquid chromatography-mass spectrometry (LC-MS/MS). TNF-α levels were measured by ELISA method.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, School of Dentistry, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Di Gangi IM, Chiandetti L, Gucciardi A, Moret V, Naturale M, Giordano G. Simultaneous quantitative determination of N(G),N(G)-dimethyl-L-arginine or asymmetric dimethylarginine and related pathway's metabolites in biological fluids by ultrahigh-performance liquid chromatography/electrospray ionization-tandem mass spectrometry. Anal Chim Acta. 2010 Sep 16;677(2):140-8. doi: 10.1016/j.aca.2010.08.011. Epub 2010 Aug 17. PMID 20837180
- [Derived] Bal I, Balci N, Sorguc C, Toygar HU, Serdar CC, Kurgan S, Serdar MA. Trimethylamine N-Oxide (TMAO) and TNF-alpha Levels in Periodontal Disease Associated With Smoking. Oral Dis. 2025 Jul;31(7):2282-2292. doi: 10.1111/odi.15262. Epub 2025 Jan 30. PMID 39887517